CLINICAL TRIAL: NCT03638466
Title: Exploratory Neuroimaging Study to Evaluate the Effect on Brain Activity of SPN-810 for Impulsive Aggression (IA) in Patients With Attention-Deficit/Hyperactivity Disorder (ADHD) in Conjunction With Standard ADHD Treatment
Brief Title: Exploratory fMRI Study on the Treatment for Impulsive Aggression in Children With ADHD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Financial decision
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 810P204
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-02

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD); Impulsive Aggression
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Magnetic Resonance Imaging; Positron-Emission Tomography; Saposins; potassium channel subfamily K member 3

STUDY DESIGN:
Intervention Model Description: A multi-center, double-blind, randomized (1:1), placebo-controlled, parallel-group, 2-arm study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High dose SPN-810 (36 mg) (Active Comparator): Subjects were randomized to receive SPN-810 18 mg twice a day twice each day with and without food, in addition to the stable dose of the optimized ADHD medication.
  Interventions: Diagnostic Test: Functional Magnetic Resonance Imaging (fMRI); Diagnostic Test: Magnetic Resonance Spectroscopy (MRS); Behavioral: Point Subtraction Aggression Paradigm (PSAP) Task; Drug: SPN-810
- Placebo (Placebo Comparator): Subjects were randomized to receive Placebo twice a day twice each day with and without food, in addition to the stable dose of the optimized ADHD medication.
  Interventions: Diagnostic Test: Functional Magnetic Resonance Imaging (fMRI); Diagnostic Test: Magnetic Resonance Spectroscopy (MRS); Behavioral: Point Subtraction Aggression Paradigm (PSAP) Task; Drug: Placebo

INTERVENTIONS:
Diagnostic Test: Functional Magnetic Resonance Imaging (fMRI) — Neural brain activity measured by fMRI
Diagnostic Test: Magnetic Resonance Spectroscopy (MRS) — Glutamate and GABA levels measured by MRS
Behavioral: Point Subtraction Aggression Paradigm (PSAP) Task — Aggression score measured by the PSAP task
Drug: SPN-810 — Treatment of SPN-810 (36 mg) on neuronal brain activity, GABA and Glutamate levels and on the aggression score
  Arms: High dose SPN-810 (36 mg)
Drug: Placebo — Treatment of placebo on neuronal brain activity, GABA and Glutamate levels and on the aggression score
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the effect of 4-week SPN-810 treatment on brain functioning in patients aged 8-12 years with ADHD and associated feature of impulsive aggression (IA). This was achieved using functional magnetic resonance imaging (fMRI) in conjunction with the point subtraction aggression paradigm (PSAP) Task, a behavioral aggression paradigm in which subjects are provoked by having money indirectly taken from them by a fictitious opponent, simulating an aggression response.

DETAILED DESCRIPTION:
Approximately 30 subjects aged 8-12 diagnosed with ADHD and associated feature of IA were recruited in this study. The PSAP is a behavioral aggression test used to evaluate behavioral response related to impulsive aggression. The task was combined with functional MRI to evaluate the change in brain activity measured as BOLD signal (blood oxygenation level-dependent) from baseline to the end of the treatment with SPN-810.

The level of neurotransmitters Glutamate and GABA were also measured using magnetic resonance spectroscopy (MRS).

Additionally, the improvement and severity in impulsive aggression behaviors were assessed using validated scales.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy male or female subjects, aged 8-12 years, inclusive, at the time of screening with primary diagnosis of ADHD and currently receiving monotherapy treatment with an optimized US Food and Drug Administration (FDA)-approved ADHD medication.
* Impulsive aggression (IA) confirmed at screening using the R-MOAS and the Vitiello Aggression Scale.

Exclusion Criteria:

* Current or lifetime diagnosis of epilepsy, major depressive disorder, bipolar disorder, schizophrenia or related disorder, personality disorder, Tourette's disorder, fetal alcohol syndrome, or psychosis not otherwise specified.
* Currently meeting DSM criteria for autism spectrum disorder, pervasive developmental disorder, obsessive-compulsive disorder, post-traumatic stress disorder.
* Known or suspected IQ <70, pregnancy, substance or alcohol abuse.
* Known history of implanted brain stimulator, vagal nerve stimulator, ventriculoperitoneal shunt, cardiac pacemaker, orthodontic braces, or implanted medication port. Visual and hearing (≥25 dB) impairment.
* Pre-existing medical or psychological conditions that preclude being in the MRI scanner (e.g., claustrophobia, morbid obesity, or marked anxiety about the procedure).

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Meridien Research aka Florida Clinical Research Center, LLC, Lakeland, Florida
  - Florida Clinical Research Center, LLC., Maitland, Florida
  - University of South Florida- Dept. of Psychiatry and Neurosciences, Tampa, Florida

REFERENCES:
- [Background] Cherek DR, Moeller FG, Schnapp W, Dougherty DM. Studies of violent and nonviolent male parolees: I. Laboratory and psychometric measurements of aggression. Biol Psychiatry. 1997 Mar 1;41(5):514-22. doi: 10.1016/s0006-3223(96)00059-5. PMID 9046983
- [Background] Bubenzer-Busch S, Herpertz-Dahlmann B, Kuzmanovic B, Gaber TJ, Helmbold K, Ullisch MG, Baurmann D, Eickhoff SB, Fink GR, Zepf FD. Neural correlates of reactive aggression in children with attention-deficit/hyperactivity disorder and comorbid disruptive behaviour disorders. Acta Psychiatr Scand. 2016 Apr;133(4):310-23. doi: 10.1111/acps.12475. Epub 2015 Aug 21. PMID 26292852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multi-center, double-blind, randomized (1:1), placebo-controlled, parallel-group, 2-arm study
Groups:
- Placebo: Subjects were randomized to receive Placebo twice each day, with or without food preferably every 12 hours, in addition to the stable dose of the optimized ADHD medication.
- High Dose SPN-810 (36 mg): Subjects were randomized to receive SPN-810 18 mg twice each day, with or without food preferably every 12 hours, in addition to the stable dose of the optimized ADHD medication.
Period: Overall Study
Arm/Group | Placebo | High Dose SPN-810 (36 mg)
Started (The number of subjects is based on the Safety Population, which included all subjects randomized and who received at least 1 dose of study drug.) | 4 | 3
Randomized Population (The Randomized Population consists of all enrolled subjects who completed the Baseline Period including imaging scans, meet the inclusion/exclusion criteria and were randomized to SPN-810 36 mg or Placebo.) | 4 | 3
Completed Population (Completed Population included all subjects randomized, who had a Baseline imaging scan (including the anatomical scan) and a valid post-treatment imaging scan.) | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 1
Not completed — Early Termination | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Population: The Randomized Population consists of all enrolled subjects who completed the Baseline Period including imaging scans, meet the inclusion/exclusion criteria and were randomized to SPN-810 36 mg or Placebo.
Groups:
- Placebo: Subjects treated with Placebo
- High Dose SPN-810 (36 mg): Subjects treated with SPN-810
- Total: Total of all reporting groups
Arm/Group | Placebo | High Dose SPN-810 (36 mg) | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 3 | 7
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.5 (1.29) | 11.3 (1.15) | 10.3 (1.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7
Vitiello Aggression Total Score [Mean (Standard Deviation); unit: units on a scale] — The Vitiello Aggression Scale is a 10-item rating scale that uses a cluster analysis to categorize aggression into two subtypes: predatory (or planned) and affective (or impulsive). The predatory score is calculated by summing up the individual scores from items 2, 5, 7, 9, and 10. The affective score is calculated by summing up the individual scores from items 1, 3, 4, 6, and 8. The total score is the difference of predatory score and affective score. Possible range of total score varies from 5 (completely predatory) to -5 (completely affective).
  units on a scale | -3.5 (1.29) | -3.7 (1.53) | -3.6 (1.27)
Retrospective-Modified Overt Aggression Scale (R-MOAS) Total Score [Mean (Standard Deviation); unit: units on a scale] — R-MOAS scale gauges the severity of aggressive behavior: the frequency of the 16 behaviors is rated over the past week in 4 areas (a-d). For each open question in each area, the parent rates the aggressive behaviors on a scale from 0 to 5 or more times. To each area corresponds a weighted category: 1(a), 4(b), 2(c) and 3(d). Therefore, the sum of each area yields a maximum weighted score of 20 (a), 120 (b), 60 (c) and 90 (c). The total score is the sum of the four area scores or 0-290, the higher the score, the more severe the aggressive behavior is.
  units on a scale | 102.5 (32.30) | 57.0 (6.00) | 83.0 (33.54)
Impulsive Aggression Measured by Clinical Global Impression - Severity Scale (CGI-S) Score [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity of Illness (CGI-S) is a single item clinician rating of clinician's assessment of a subject's global functioning prior to administration of a study medication. CGI-S was evaluated by the Investigator on a 7- point scale with 1=Normal, 2=Borderline ill, 3=Mildly ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, and 7=Extremely ill.
  units on a scale | 5.8 (0.96) | 5.0 (1.41) | 5.5 (1.05)

OUTCOME MEASURES:

1. Primary Outcome: Aggression-related Change in the Whole Brain in BOLD (Blood Oxygenation Level-dependent) Signal fMRI Contrast in Response to the PSAP Task
Description: The primary endpoint was the aggression-related change in the whole brain in BOLD signal fMRI contrast in response to the PSAP task. BOLD fMRI contrast (neural activation) investigates brain activity by measuring the change in blood oxygenation. Change in brain activity was measured by a change in BOLD response in brain regions during the aggressive response relative to the monetary response, where the aggression was defined as the number of Option 2 presses (aggressive response) divided by the total number of button presses and the number of provocations. Change of aggression-related MRI signal was acquired at baseline and 4 weeks after SPN-810 treatment. A positive number represents an increase in activity. Region of interest is described by the location of the peak value and described by Montreal Neurological Institute (MNI) X, Y, Z coordinates. Data represent the post-treatment minus baseline change in BOLD contrast Aggressive Response> Monetary Response.
Time Frame: Baseline/Visit 2 (Day -5) to Visit 5 (Day 28) for a total of 4 weeks.
Population: Completed population included all subjects randomized, who had a Baseline imaging scan (including the anatomical scan) and post-treatment imaging scans.
Measure: Mean (95% Confidence Interval); unit: Voxels
Groups:
- SPN-810 (36 mg) > Placebo: Increase over placebo BOLD response in subjects treated with high dose of SPN-810
- Placebo > SPN-810 (36 mg): Increase over high dose of SPN-810 BOLD response in subjects treated with placebo
Arm/Group | SPN-810 (36 mg) > Placebo | Placebo > SPN-810 (36 mg)
Number analyzed (Participants) | 2 | 4
Voxels
  Inferior Occipital Gyrus/Cerebellum: Montreal Neurological Institute coordinates -29.5, 62.5, -4.5 | 353 [310.6 to 395.4] | 0 [0 to 0]
  Right Fusiform Gyrus/Inferior Occipital Cortex: Montreal Neurological Institute 32.5, 52.5, 23.5 | 258 [223.1 to 292.9] | 0 [0 to 0]
  Left Angular Gyrus (WM): Montreal Neurological Institute coordinates 4.5, 84.5, 35.5 | 173 [145.2 to 200.8] | 0 [0 to 0]
  Left Cuneus: Montreal Neurological Institute coordinates -23.5, 96.5, 5.5 | 145 [124.6 to 165.4] | 0 [0 to 0]
  Right Middle Occipital Gyrus: Montreal Neurological Institute coordinates -1.5, 64.5, 57.5 | 133 [114.2 to 151.8] | 0 [0 to 0]
  Medial Precuneus: Montreal Neurological Institute coordinates -33.5, 34.5, 47.5 | 128 [111.3 to 144.7] | 0 [0 to 0]
  Right Postcentral Gyrus: Montreal Neurological Institute coordinates -29.5, 62.5, -4.5 | 110 [95.1 to 124.9] | 0 [0 to 0]
  Superior Medial Frontal Gyrus: Montreal Neurological Institute coordinates 2.5, -47.5, 39.5 | 0 [0 to 0] | 329 [288.6 to 369.4]
  Right Cerebellum: Montreal Neurological Institute coordinates: -35.5, 72.5, -40.5 | 0 [0 to 0] | 175 [145.2 to 204.8]
  Right Superior/Middle Frontal Gyrus: Montreal Neurological Institute coordinates -37.5, -33.5, 33.5 | 0 [0 to 0] | 164 [136.2 to 191.8]
  Right Insula Montreal Neurological Institute coordinates -39.5, -13.5, -0.5 | 0 [0 to 0] | 140 [116.4 to 163.6]
  Right Inferior Temporal Gyrus: Montreal Neurological Institute coordinates -41.5, -7.5, -46.5 | 0 [0 to 0] | 145 [124.6 to 165.4]
  Left Postcentral Gyrus: Montreal Neurological Institute coordinates 30.5, 30.5, 51.5 | 0 [0 to 0] | 110 [95.1 to 124.9]

2. Primary Outcome: Provocation Event - Related Change in the Whole Brain in BOLD Signal fMRI Contrast in Response to the PSAP Task
Description: BOLD (blood oxygenation level-dependent) fMRI contrast (neural activation) investigates brain activity by measuring the change in blood oxygenation. It was collected during the PSAP behavioral task while playing the game: the participants play a computer game in which they can steal points (simulating an aggressive behavior) or have points stolen by the opponent (provocation event) by pressing Option 1, 2 or 3 on a keypad a set number of times to achieve a specific outcome. A positive number represents an increase in activity. The region of interest is described by the location of the peak value within that cluster and described by Montreal Neurological Institute (MNI) X, Y, and Z coordinates. Data represent the post-treatment minus baseline change in BOLD contrast Provocation Event >Monetary Response.
Time Frame: Baseline/Visit 2 (Day -5) to Visit 5 (Day 28) for a total of 4 weeks.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Voxels
Arm/Group | SPN-810 (36 mg) > Placebo | Placebo > SPN-810 (36 mg)
Number analyzed (Participants) | 2 | 4
Voxels
  Right Postcentral Gyrus: Montreal Neurological Institute coordinates: -31.5, 30.5, 43.5 | 318 [276.3 to 359.7] | 0 [0 to 0]
  Left Middle/Inferior Temporal Gyrus: Montreal Neurological Institute coordinates 52.5, 16.5, -24.5 | 137 [117.5 to 156.5] | 0 [0 to 0]
  Medial Cerebellum: Montreal Neurological Institute coordinates: 12.5, 50.5 -32.5 | 0 [0 to 0] | 123 [104.1 to 141.9]
  Left Inferior Frontal Gyrus: Montreal Neurological Institute coordinates: 42.5, -15.5, 19.5 | 0 [0 to 0] | 122 [105.0 to 139.0]
  Right Cerebellum: Montreal Neurological Institute coordinates: -23.5, 70.5, -24.5 | 0 [0 to 0] | 109 [94.4 to 123.6]

3. Primary Outcome: Effect of SPN-810 on the Aggressions Score
Description: The Point Subtraction Aggression Paradigm (PSAP) is a behavioral aggression paradigm consisting of a computer game in which each participant plays against a computer to earn points. The subject can steal points (i.e., aggressive behavior) or have points stolen by the opponent (i.e., provocation). The subject can press 1 of 3 buttons on a keypad a set number of times. By pressing the button for Option 1, 100 times, the subject will earn a point; pressing the button for Option 2, 20 consecutive times is the "aggression" action that results in stealing a point from the opponent; pressing Option 3, 20 times protects the subject from the opponent's attempt to steal points (i.e., money). The aggression score is averaged across two sessions and calculated as the number of Option 2 button presses divided by the sum of total button presses and the number of provocation events received, with a range minimum = 1, maximum = 143. The higher scores reflect increased aggression.
Time Frame: Baseline/Visit 2 (Day -5) to Visit 5 (Day 28) for a total of 4 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- High Dose SPN-810 (36 mg): Subjects treated with high dose of SPN-810
Arm/Group | Placebo | High Dose SPN-810 (36 mg)
Number analyzed (Participants) | 4 | 2
score on a scale
  Baseline/Visit 2 | 8.43 (9.22) | 10.23 (6.21)
  Visit 5 | 9.26 (5.50) | 4.02 (2.60)

4. Secondary Outcome: Effect of SPN-810 on GABA and Glutamate Levels Using Magnetic Resonance Spectroscopy (MRS)
Description: GABA and Glutamate concentrations (mM) were measured in the anterior cingulate cortex using magnetic resonance spectroscopy (MRS). Data represent the change from Baseline (Visit 2) to Visit 5.
Time Frame: Baseline/Visit 2 (Day -5) to Visit 5 (Day 28) for a total of 4 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mM
Groups:
- High Dose of SPN-810 (36 mg): Subjects treated with high dose of SPN-810
Arm/Group | Placebo | High Dose of SPN-810 (36 mg)
Number analyzed (Participants) | 4 | 2
mM
  GABA (mM) | 0.79 (0.26) | 0.75 (0.67)
  Glutamate (mM) | 0.78 (2.44) | 0.23 (1.91)

5. Other Pre Specified Outcome: Effect of SPN-810 on Impulsive Aggression Measured by the Clinical Global Impression-Severity (CGI-S) Scale
Description: The Clinical Global Impression - Severity of Illness (CGI-S) is a single item clinician rating of clinician's assessment of the severity of IA behaviors. CGI-S was evaluated by the Investigator on a 7- point scale with 1=Normal, 2=Borderline ill, 3=Mildly ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, and 7=Extremely ill. Data represent the change between Baseline (Visit 1/Day -30) and two time points: Visit 4 (Day 21) and Visit 6 (Day 35).
Time Frame: From Visit 1 (Day -30) to two time points: Visit 4 (Day 21) and Visit 6 (Day 35).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- High Dose SPN-810: Subjects treated with 36 mg SPN-810
Arm/Group | Placebo | High Dose SPN-810
Number analyzed (Participants) | 4 | 2
score on a scale
  Visit 4 | -1.25 (1.5) | -1.5 (2.12)
  Visit 6 | -2.25 (1.5) | -1.5 (2.12)

6. Other Pre Specified Outcome: Effect of SPN-810 on Impulsive Aggression Measured by the Clinical Global Impression-Improvement (CGI-I) Scale
Description: The Clinical Global Impression - Improvement Scale (CGI-I) is an assessment of how much the patient's illness has improved or worsened relative to a baseline state at the beginning of treatment.
  CGI-I was evaluated by the Investigator on a 7-point scale with 1=very much improved, 2= much improved, 3= minimally improved, 4= no change, 5= minimally worse, 6= much worse, 7= very much worse.
Time Frame: Visit 4 (Day 21) and Visit 6 (Day 35), for a total of 2 weeks.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Subjects will be treated with a matching Placebo
- High Dose of SPN-810 (36 mg): Subjects treated with a high dose of SPN-810
Arm/Group | Placebo | High Dose of SPN-810 (36 mg)
Number analyzed (Participants) | 4 | 2
score on a scale
  Visit 4 | 2.3 (1.26) | 1.5 (0.71)
  Visit 6 | 2.3 (1.26) | 1.0 (0.0)

7. Other Pre Specified Outcome: Effect of SPN-810 on the Retrospective-Modified Overt Aggression Scale (R-MOAS) Score
Description: R-MOAS scale gauges the severity of aggressive behavior: the frequency of the 16 behaviors is rated over the past week in 4 areas (a-d). For each open question in each area, the parent rates the aggressive behaviors on a scale from 0 to 5 or more times. To each area corresponds a weighted category: 1(a), 4(b), 2(c) and 3(d). Therefore, the sum of each area yields a maximum weighted score of 20 (a), 120 (b), 60 (c) and 90 (c). The total score is the sum of the four area scores or 0-290, the higher the score, the more severe the aggressive behavior is. Data represent the change from baseline at each visit.
Time Frame: Visit 1 (Day -30) to Visit 4 (Day 21) and Visit 6 (Day 35).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | High Dose SPN-810 (36 mg)
Number analyzed (Participants) | 4 | 2
score on a scale
  Visit 4 | -52.0 (30.23) | -43.0 (2.83)
  Visit 6 | -61.0 (18.81) | -39.5 (24.75)

ADVERSE EVENTS:
Time Frame: Visit 3 (Day 1) to Visit 6 (Week5)-End of Study, a total of 5 weeks
Description: Adverse events reporting pertains to the Safety Population which included all subjects randomized and who received at least 1 dose of study drug.
Arm/Group | Placebo | High Dose SPN-810
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 2/4 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4) | High Dose SPN-810 (N=3)
Fatigue (General disorders) | 1 | 0
Decrease appetite (Metabolism and nutrition disorders) | 2 | 0
Blood Prolactin Increased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT03638466/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT03638466/SAP_001.pdf